CLINICAL TRIAL: NCT04356157
Title: WeMen! Improving Women's Access to Healthcare System Through Men's Inclusion
Acronym: WEMEN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Rome Tor Vergata (Other)
Collaborators: Scuola Superiore Sant'Anna di Pisa (Other); Comunità di S.Egidio ACAP Onlus (Unknown); Ministero degli Affari Esteri Italia (Unknown)
Responsible Party: Principal Investigator, Leonardo Palombi, Full Professor, University of Rome Tor Vergata
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: AID-011587/08/05
Record Dates: First submitted 2020-04-10; First posted 2020-04-22 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: HIV
Keywords: Retention; Adherence; Male involvement; HIV; Interventions; Malawi

STUDY DESIGN:
Intervention Model Description: The three interventions to be implemented and evaluated in the research plan are designed to assess the involvement of MI at individual level, interpersonal/network, community-level, Health System and structural level according to ecological model.
  The study is articulated in three phases: pre-intervention, intervention and post-intervention analyses. In the pre-intervention analysis, the baseline situation of the three participating centres will be evaluated. The aim of this phase is to set a starting point in order to weigh the relative effect of each intervention to be studied. In each clinical centre baseline data will be collected. In order to evaluate the effect of the interventions, the same indicators will be measured in pre-and in post-intervention phase. The enrollment of participants will be consecutively based on the order of patient appointments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Special day (Other): The special day takes place with an extraordinary opening of the clinical centre once a month on a pre-festive day (Saturday). During this day, access will be reserved exclusively for men, including those who are not on treatment for HIV. The centre will offer free health promotion services to all participants.
  Interventions: Behavioral: Behavioural change interventions
- Male Champions (Other): The "male champion" is a figure present in a few settings which carries out home visits with men and couples and follows up with men who did not accompany their partners to Antenatal Care visits. Usually, this role is covered by the female Expert Clients, namely HIV+ patients working in the organization as volunteers after appropriate training. Some men among patients who are on treatment will be identified and trained to cover this role.
  Interventions: Behavioral: Behavioural change interventions
- Nudge (Other): The intervention based on the use of incentives (nudge) to men who follow the prevention and treatment program aims to evaluate whether this action is effective in guiding behaviour change towards the test, treatment, involvement and adherence to therapy approach.
  Interventions: Behavioral: Behavioural change interventions
- No intervention (Other): No intervention will be carried out in a center.
  Interventions: Behavioral: Behavioural change interventions

INTERVENTIONS:
Behavioral: Behavioural change interventions — The study evaluates three different interventions aimed at improving adherence and retention to Anti Retroviral therapy among HIV positive women through engagement with their life partner. The interventions are 1) opening the facility once a month, only for men, "special day"; 2) testing peer-to-peer counselling among men, "male champions"; 3) providing incentive to all women accompanied by their partners at the facility, "nudge" or "incentive".

SUMMARY:
Background: More than two-thirds of people living with HIV live in Sub-Saharan Africa, where the HIV prevalence in the adult population (aged 15-49) is 3.9%.

In these countries a critical issue is represented by low level of adherence to treatment particularly in HIV positive pregnant women. Among the causes, the lack of male partner involvement represents a significant criticality. This issue emerge in Malawi, one of the countries with the highest prevalence of HIV in the world: 9.2% of the adult population living with HIV in 2018.

Objective: to assess three different interventions aimed at improving adherence and retention to Anti Retroviral therapy among HIV positive women through engagement with their life partner in four Malawian healthcare centres.

Methods: The prospective, controlled before-and-after study is articulated in three phases (total 24 months): pre-intervention, intervention and post-intervention analyses. The number of selected clinical centres is limited to four, one for each intervention plus a centre where no intervention will be performed (control arm). The interventions are 1) opening the facility on Saturday a month, only for men, defined "special day"; 2) peer-to-peer counselling among men, "male champions"; 3) providing incentive to all women accompanied by their partners at the facility, "nudge" (note1).

The primary outcome of the study is the evaluation of the variations in retention in care and women's adherence to therapeutic protocols; the intermediate outcome is the assessment of the variations in Male Involvement (MI).

The level of MI in the health of female partners (intermediate outcome) will be evaluated through a questionnaire administered at baseline and in the post-intervention phase. Data will be collected at the clinical centres and will be stored in two electronic databases.

Results: Analysis of data collected in the four centres during the pre-intervention phase is on-going as the enrolment is stopped 31st March 2020. Total patients enrolled are 452 (133 Namandanje: 133, Kapeni: 78, Kapire: 75, Balaka: 166). Meantime, several meetings are performed in the centres to organize the intervention phase.

Conclusions: The study will identified the better intervention to involve male partners in women's health according to an approach based on a broad spectrum of behaviours.

- Note1: the reason of the incentive is not reward the participation in the study but is the main activity of the intervention assessed. The intervention consist in giving an incentive. For this reason is not recommendable to eliminate this information as requested by the reviewer.

DETAILED DESCRIPTION:
The design is a prospective controlled study, that is suitable for the evaluation of promising interventions to improve male involvement and enhance maternal adherence to HIV PMTCT.

For this study, we adopted a framework based on the ecological model adapted by Kaufman et al to health behaviors in HIV prevention.

According to the ecological model, many factors affect male involvement in women's health care processes at different levels. In this study, we focused on individual level, interpersonal and network (eg, family and peers), community, health system (health facility level), and structural level (eg, access to transportation).

The aim of the study is to evaluate 3 different interventions aimed at improving adherence and retention to Anti Retroviral therapy among HIV-positive women through engagement with their life partner. The interventions are (1) testing peer-to-peer counseling and community-level health education sessions delivered by men, male champions; (2) opening the facility once a month, only for men, special day; and (3) providing incentive to all women accompanied by their partners at the facility, nudge or incentive (note1).

* Intervention 1 (Male Champions) will act at the community level, providing educational interventions that are aimed at territorial communities and religious groups.
* Intervention 2 (Special Day) will act at the health system level delivering activities based on health facilities that are aimed at reshaping the clinic as male-friendly.
* Intervention 3 will also act at the structural level by providing incentives to support the cost of transportation and other costs that reduce a male partner's ability to access the service (note1).

The study has 3 phases: preintervention (baseline), intervention, and postintervention analyses, as shown in Figure 2.

In the preintervention analysis, the baseline situation of the 3 participating centers will be evaluated. The aim of this phase is to set a starting point to weigh the relative effect of each intervention to be studied. For that purpose, baseline data of each study site will be collected. To evaluate the effect of the interventions, the same indicators will be measured during the pre- and postintervention phases, as described above. The preintervention phase will last 9 months. During this period, data will be collected at each site and included in a database.

Given the limited resources available for the study and the practical difficulties related to the disadvantaged context in which the study was conducted, sample size calculations and criteria for assigning interventions were based on a pragmatic approach. The number of selected clusters is limited to 4, one for each intervention plus a cluster where no intervention will be performed as a control arm. The number of participants enrolled for data collection is given by the number of patients attending the selected clinical centers during the pre- and postintervention phases. Therefore, the main unit of analysis of the study is the cluster, which is the clinical center. Thus, the interventions will target each health facility.

The following criteria were followed to select the 4 centers included in the intervention:

1. The centers represented the Malawian population. As Malawi is a country where 83% of the population resides in rural or semirural environments, rural clinics were selected.
2. Centers that only provided maternal services were excluded because it was not possible to use a male-friendly approach in a center that is designed to accommodate only women.
3. The remaining centers with the highest number of female patients were selected. The special day intervention was assigned to the center of Balaka (Balaka district). At this site, health care staff are available to offer the planned services. The male champion intervention was assigned to the Kapire center (Machinga district), where there are patients available to engage themselves as male champions who have sufficient levels of education necessary to perform the task assigned to them and communicate with the researchers. The nudge intervention was assigned to the Kapeni center (Blantyre district), where the number of women being treated was consistent with the available budget necessary for the provision of noneconomic incentives (note1).

Although the unit of analysis is the clinical center, and therefore all patients who are referred, the study focuses on the population of adult females and the influence of male partners on the health practices of women. Therefore, data will be collected from this specific population. Eligibility criteria for women included the following: being HIV positive; inclusion in an HIV/AIDS prevention and treatment program; aged 18 years or older; and living at home with a male partner.

The enrollment of participants will be consecutively based on the order of patient appointments. Recruitment will be entrusted to doctors and clinical officers responsible for the medical visits of women participating in HIV treatment programs, who interact with patients during every visit to the clinical center. All women who met the eligibility criteria and agreed to participate in the study will be enrolled. Recruitment will be conducted before the medical examination: the software used for patient management reports to the clinician whether patients aged less than 18 years are enrolled, allowing the clinician to check entry criteria and invite eligible participants for study participation with the provision of informed consent.

Data will be collected at the clinical centers and will be stored in 2 electronic databases managed through 2 different types of software:

1. Clinical and medical service data are routinely collected through an electronic DREAM program health record software used routinely at the clinical centers named DREAM_S.
2. Data on health behaviors reported by patients who participate in the study will be collected through the software created specifically for the study, also respecting rules for patient privacy and data security.

In the preintervention phase, data will be collected at the medical visit immediately after the enrollment visit to evaluate the partner's acceptance of the invitation to come to the clinical center for testing and counseling in the company of the patient. In the postintervention phase, data will be collected 2 months from enrollment to allow for a wash-out period where the effects of the interventions would be expressed.

The interventions will be implemented according to standard clinical practices in Malawi with some modifications based on the international experiences described in the literature.

1. The male champion is a figure present in a few settings that conducts home visits with men and couples and follows up with men who did not accompany their partners to Ante-Natal Care (ANC) visits. Usually, this role is covered by the female expert clients, namely HIV-positive patients working in the organization as volunteers after appropriate training. Some men among patients who are receiving treatment will be identified and trained to cover this role. The intervention called male champion aims to change the beliefs and attitudes of men, not intervening directly on individuals but upon entire communities and particularly involving community leaders.
2. The special day is a practice that is becoming increasingly common to facilitate access to health facilities by vulnerable groups such as adolescents. In this study, we target men. The special day takes place with an extraordinary opening of the clinical center once a month on a pre-festive day (Saturday). During this day, access will be reserved exclusively for men, including those who are not on treatment for HIV. The center will offer free health promotion services to all participants. This intervention aims to remove the attitude linked to beliefs regarding masculinity, in which the male partners see access to health centers as an activity suitable only for women. The special day aims to make the clinical center more male-friendly and therefore attempts to overcome the social pressure that pushes men to have only sporadic attendance.
3. The intervention based on the use of incentives (nudge) to men who follow the prevention and treatment program aims to evaluate whether this action is effective in guiding behavior change toward the test, treatment, involvement, and adherence to therapy approach. The intervention defined as nudge aims to remove the obstacles of a structural or a material nature, therefore it supports the costs related to transportation to health care facilities and time taken away from work through a noneconomic incentive (note1).

The educational tools developed for these interventions are based on standards adopted in the country for couples counseling on HIV/AIDS. To these standard guidelines, messages were added to initiate a reflective discussion of stereotypes and false beliefs related to the idea of masculinity in the Malawian culture. All staff involved in the delivery of these interventions were provided with a guide (included in Multimedia Appendix 1) on the contents to be delivered. They also participated in a one-day training of the themes of the project. The guide was developed by study investigators and Malawian health care staff. The guide was based on tools developed and applied in other contexts with the purpose of increasing men's access to health care services and to reduce stereotypes and gender-based violence. It was also based on the ecological model.

The educational content will be delivered using 3 different approaches. The special day arm will address the community in the catchment area of the clinical center, but the intervention will take place at the facility level. Through visibility activities such as leaflet distributions or information campaigns with audio messages, men living in the communities surrounding the treatment center will be invited to an extraordinary opening day at the center dedicated only to men. During the special day, the center's clinical staff will offer basic health care services such as HIV testing and counseling, blood pressure measurement and counseling on cardiovascular disease, blood glucose measurement and counseling on diabetes, and nutritional evaluation and counseling. During the morning, group educational activities led by male community health care workers together with the doctors of the center and 2 educational sessions using drama techniques will be conducted. In the male champions arm, the intervention will be conducted at the level of regional and religious communities, with group educational sessions and use of the male champions. Male champions will be selected from patients receiving treatment for HIV for more than a year at the local DREAM centers. The educational sessions, based on an interactive approach with questions and answers both from the audience and the male champions, will last between 30 min to an hour. The male champion will be allowed to prolong the intervention if the audience requests it. Meetings will be planned and implemented in communities where at least five patients who receive treatment at DREAM centers reside, including religious communities in those regions. In the nudge arm, the intervention will be directed to individuals or to male partners of female patients being treated at DREAM centers. Women who agree to participate in the study will be asked to invite their male partners to the center for a health education session, and male partners who agree to participate will receive an incentive for attending the service in the form of a food package (note1). At the second visit, the couple will be given a health education session based on educational materials prepared for the study.

- Note1: the reason of the incentive is not reward the participation in the study but is the main activity of the intervention assessed. The intervention consist in giving an incentive. For this reason is not recommendable to eliminate this information as requested by the reviewer.

ELIGIBILITY:
Inclusion Criteria:

* Being HIV positive
* Inclusion in an HIV/AIDS prevention and treatment program
* Age of 18 years or older
* Living at home with a male partner

Exclusion Criteria:

* No HIV positive
* No included in a HIV/AIDS prevention and treatment program
* Under 18 years old
* No partner living at home

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Retention in care and adherence to treatment | 2 years
  Retention in care will be measured as the cumulative proportion of dropouts from the treatment program at 6 months, 1 year, and 2 years (excluding patients transferred to another centre or those who died). Adherence will be measured through the following indicators: (1) The cumulative proportion of medical appointments missed in a month period in the centre; (2) the cumulative proportion of appointments for drug delivery missed in a month period in the centre; (3) the cumulative proportion of women who suppressed viral load; (4) the cumulative proportion of women with a suppressed viral load that have a re-bound in viremia.

SECONDARY OUTCOMES:
Male Involvement - Proportion of women accompanied by partners | 2 years
  Proportion of women accompanied by partners at the facility after receiving an invitation card;
Male Involvement 2 - Proportion of men accepting HIV testing and counselling | 2 years
  Proportion of men accepting HIV testing and counselling (if not yet received in the last 6 months)
Male Involvement 3 - Score scale of MI in health practices reported from female partners | 2 years
  level of partner's involvement in the care process measured through a score scale based on health practices reported by the female partners
Male Involvement 4 - Score scale of Gender Based Violence reported from female partner | 2 years
  Level of gender-based violence in the family measured through a score scale based on the violent/negative practices reported by female partners.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Palombi, MD, PhD, Principal Investigator — Università Tor Vergata Roma
Locations (4):
- Malawi (4):
  - Balaka DREAM centre, Balaka
  - Kapeni DREAM centre, Blantyre
  - Namandanje DREAM centre, Machinga
  - Kapire DREAM centre, Mangochi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Triulzi I, Palla I, Ciccacci F, Orlando S, Palombi L, Turchetti G. The effectiveness of interventions to involve men living with HIV positive pregnant women in low-income countries: a systematic review of the literature. BMC Health Serv Res. 2019 Dec 9;19(1):943. doi: 10.1186/s12913-019-4689-6. PMID 31815620
- [Background] Aliyu MH, Sam-Agudu NA, Shenoi S, Goga AE, Ramraj T, Vermund SH, Audet CM. Increasing male engagement in the prevention of vertical transmission of HIV: what works in sub-Saharan Africa? BMJ. 2019 Jun 6;365:l1965. doi: 10.1136/bmj.l1965. PMID 31171558
- [Background] Takah NF, Kennedy ITR, Johnman C. The impact of approaches in improving male partner involvement in the prevention of mother-to-child transmission of HIV on the uptake of maternal antiretroviral therapy among HIV-seropositive pregnant women in sub-Saharan Africa: a systematic review and meta-analysis. BMJ Open. 2017 Nov 25;7(11):e018207. doi: 10.1136/bmjopen-2017-018207. PMID 29175889
- [Background] Mancinelli S, Nielsen-Saines K, Germano P, Guidotti G, Buonomo E, Scarcella P, Lunghi R, Sangare H, Orlando S, Liotta G, Marazzi MC, Palombi L. Who will be lost? Identifying patients at risk of loss to follow-up in Malawi. The DREAM Program Experience. HIV Med. 2017 Sep;18(8):573-579. doi: 10.1111/hiv.12492. Epub 2017 Feb 2. PMID 28150466
- [Background] Matseke MG, Ruiter RAC, Rodriguez VJ, Peltzer K, Setswe G, Sifunda S. Factors Associated with Male Partner Involvement in Programs for the Prevention of Mother-to-Child Transmission of HIV in Rural South Africa. Int J Environ Res Public Health. 2017 Nov 1;14(11):1333. doi: 10.3390/ijerph14111333. PMID 29104275
- [Background] Kaufman MR, Cornish F, Zimmerman RS, Johnson BT. Health behavior change models for HIV prevention and AIDS care: practical recommendations for a multi-level approach. J Acquir Immune Defic Syndr. 2014 Aug 15;66 Suppl 3(Suppl 3):S250-8. doi: 10.1097/QAI.0000000000000236. PMID 25007194
- See also: DREAM programme website — https://www.dream-health.org